CLINICAL TRIAL: NCT01613677
Title: Phase II, Open Label, Non-randomized, Trial of BKM120 as Palliative Treatment for Metastatic or Locally Advanced Cervical Cancer After Failure to Platinum Based Regimen
Brief Title: Phase II, Open Label, Non-randomized, Trial of BKM120 for Metastatic or Locally Advanced Cervical Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBKM120ZBR01
Record Dates: First submitted 2012-06-05; First posted 2012-06-07 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2016-02

CONDITIONS: Treatment for Metastatic or Locally Advanced Cervical Cancer
Keywords: advanced cervical cancer, BKM 120, progression free survival
MeSH Terms: interventions — NVP-BKM120

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BKM120 (Experimental)
  Interventions: Drug: BKM120

INTERVENTIONS:
Drug: BKM120

SUMMARY:
This is a single arm open label phase II trial to evaluate the oral daily use of BKM 120 in patients with recurrent unresectable or metastatic cervical cancer after palliative cisplatin based regimen failure.

A complete treatment cycle is defined as a 28 days period.

DETAILED DESCRIPTION:
Inclusion and exclusion criteria should be assessed in the pretreatment visit and the informed consent must be taken before treatment assignment. The diagnosis and extent of disease, the medical history, and the current medical condition should be recorded by the investigator in a pretreatment visit. Adverse events will be recorded including type, severity, graded by CTCAE V 3.0, seriousness and potential relation to the investigational drug.

The efficacy assessment will be done by MRI and recorded in the patients' clinical chart. Tumor dimension assessments will be performed at baseline through abdominal/pelvic magnetic resonance imaging, to be repeated in 3 months intervals and evaluated according RECIST criteria. The first cohort, composed by the 06 first patients, will undergo a separate positron-emission tomography (PET-CT) evaluation at baseline and 90 days apart.

Laboratory tests (hematology, blood chemistry), ECG and physical examination will be done on every visit.

Drug pharmacokinetics will not be assessed in this study. For the screening Baseline periods, see chart attached The treatment will be continued until progressive disease or intolerable toxicity

ELIGIBILITY:
Inclusion Criteria:

* Patient has provided a signed Informed Consent Form (ICF) obtained prior to any screening procedure.
* Female 18 years of age or older.
* Histologically or cytologically confirmed recurrent unresectable or metastatic cervix squamous-cell carcinoma.
* ECOG performance status 0-2
* Adequate renal, hepatic and hematologic function:

  * ANC ≥1250/mm3;
  * Platelet count ≥100,000/mm3;
  * Hemoglobin ≥ 9.0 g/dL
  * Creatinine ≤1.5X upper limits of normal or 24 hrs clearance ≥55ml/min;
  * Serum bilirubin within normal range (or ≤ 1.5 x ULN if liver metastases are present; or total bilirubin ≤ 3.0 x ULN with direct bilirubin within normal range in patients with well documented Gilbert Syndrome)
  * SGOT, SGPT ≤ 1.5 X upper limits of normal if no liver metastasis present;
  * SGOT, SGPT, alkaline phosphatase ≤ 3 X upper limits of normal if liver metastasis present;
* Measurable disease by magnetic resonance imaging according to RECIST criteria.
* Willingness and capacity in understand and comply with all of the trial planned procedures, including periodic medical visits, treatment plans and laboratory tests.
* Negative serum pregnancy test during screening and negative urinary test for pregnancy within 48 hours before starting study treatment in women with childbearing potential

Exclusion Criteria:

* Previous use of a PI3K inhibitor.
* Brain or spinal cord compressive metastasis. Patients with appropriately treated brain or spinal metastasis and neurologically stable for at least 4 weeks can be included at discretion of investigator.
* Concurrent malignancy other than non-melanoma skin cancer.
* Concurrent clinical condition impeditive to be part of the study at the judgment of the investigator.
* Patient has any of the following mood disorders as judged by the Investigator or a Psychiatrist, or meets the cut-off score of ≥ 10 in the PHQ-9 or a cut-off of ≥ 15 in the GAD-7 mood scale, respectively, or selects a positive response of '1, 2, or 3' to question number 9 regarding potential for suicidal thoughts ideation in the PHQ-9 (independent of the total score of the PHQ-9):

  * Medically documented history of or active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, or homicidal ideation (immediate risk of doing harm to others)
  * ≥ CTCAE grade 3 anxiety
* Patients with acute or chronic liver, renal disease or pancreatitis.
* Patients with diarrhea ≥ CTCAE grade 2.
* Any of the following concurrent severe and/or uncontrolled medical conditions which could compromise participation in the study:

  * ST depression or elevation of ≥ 1.5 mm in 2 or more leads;
  * Congenital long QT syndrome;
  * History or presence of sustained ventricular arrhythmias or atrial fibrillation;
  * Clinically significant resting bradycardia (< 50 beats per minutes);
  * QTc > 480 msec on screening ECG;
  * Complete left bundle branch block;
  * Right bundle branch block + left anterior hemi block (bifascicular block) ;
  * Unstable angina pectoris ≤ 6 months prior to starting study drug;
  * Acute myocardial infarction ≤ 6 months prior to starting study drug;
  * Other clinically significant heart disease such as congestive heart failure requiring treatment (NYHA Class III or IV) or uncontrolled hypertension;
* Patients with clinical manifestation of diabetes mellitus (i.e. treated and/or with clinical signs) or steroid-induced diabetes mellitus or uncontrolled diabetes (Fasting glucose >120 mg/dL (HbA1c >8%).
* Other concurrent severe and/or uncontrolled concomitant medical conditions (e.g., active or uncontrolled infection) that could cause unacceptable safety risks or compromise compliance with the protocol.
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of BKM120 (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
* Patients who have received corticosteroids ≤ 2 weeks prior to starting study drug.
* Patient is currently being treated with drugs known to be moderate and strong inhibitors or inducers of isoenzyme CYP3A, and the treatment cannot be discontinued or switched to a different medication prior to starting study drug. Please refer to Table 5-8 for a list of prohibited CYP3A4 inhibitors and inducers.
* Employing an effective method of birth control. (Women of child-bearing potential, defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months (i.e., who has had menses any time in the preceding 12 consecutive months),
* must have a negative serum pregnancy test during screening and negative urinary test for pregnancy within 48 hours before starting study treatment in women with childbearing potential).
* Known diagnosis of human immunodeficiency virus (HIV) infection.
* Patient is unable or unwilling to abide by the study protocol or cooperate fully with the investigator.
* Patient has received pelvic and/or para-aortic radiotherapy ≤ 28 days prior to enrollment in this study or has not recovered from side effects of such therapy at the time of initiation of screening procedures
* MRI study - additional exclusions to consider for an MRI study

  * Cardiac pacemaker
  * Ferromagnetic metal implants other than those approved as safe for use in MR scanners (Example: some types of aneurysm clips, schrapnel)
  * Claustrophobia
  * Obesity (exceeding the equipment limits)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-11; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Toxicity profile by recording the frequency and severity of adverse events associated to the use of daily oral BKM 120 as assessed by NCI CTCAE v. 3.0 | 18 months

SECONDARY OUTCOMES:
Clinical benefit [complete response (CR), partial response (PR) rate and stable disease] according to RECIST criteria. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Biociências SA - Brazil, Study Director — Novartis
Locations (1):
- Novartis Investigative Site, Rio de Janiero, Rio de Janeiro, Brazil